CLINICAL TRIAL: NCT02929459
Title: Effects of Oral Riboflavin Supplementation on the Growth of Faecalibacterium Prausnitzii and the Impact on the Gut Microbiota: A Randomized, Double-blind, Placebo-controlled Human Intervention Trial
Brief Title: Effects of Riboflavin on Faecalibacterium Prausnitzii and the Gut Microbiota
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RiboGut2015
Record Dates: First submitted 2016-10-06; First posted 2016-10-11 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Gut Microbiota
Keywords: Gut Microbiota; Riboflavin; Vitamin B2; oGTT; Faecalibacterium prausnitzii
MeSH Terms: interventions — Riboflavin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Riboflavin Dose 1 (Experimental): 100 mg Riboflavin (one capsule) per day for 2 weeks
  Interventions: Dietary Supplement: Riboflavin Dose 1
- Riboflavin Dose 2 (Experimental): 50 mg Riboflavin (one capsule) per day for 2 weeks
  Interventions: Dietary Supplement: Riboflavin Dose 2
- Placebo (Placebo Comparator): 100 mg starch plus 0,5% silica (one capsule) per day for 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Riboflavin Dose 1
  Other Names: Vitamin B2
  Arms: Riboflavin Dose 1
Dietary Supplement: Riboflavin Dose 2
  Other Names: Vitamin B2
  Arms: Riboflavin Dose 2
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate comprehensively the effect of riboflavin supplementation on the abundance of F. prausnitzii and on other members of the gut microbiota in faeces of healthy volunteers. Additionally it will be assessed whether riboflavin supplementation affects the abundance of potentially pathogenic bacteria such as adherent invasive E. coli (AIEC). Finally, the effect of riboflavin supplementation on the production of Short Chain Fatty Acids, the release of gut hormones and potential changes in glucose homeostasis and appetite perception will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females, age 20 - 60 years
* Participant is willing to stick to his/her normal habitual diet excluding consumption of any unusual high energy-rich or fat-rich meals or prolonged fasting, etc. throughout the study period
* Participant is willing to maintain his/her habitual physical activity patterns throughout the study period
* Participant has been stable in body-weight within the last 6 months
* Participant has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the investigator on the basis of medical history and routine laboratory test results
* Participant has a body mass index (BMI) of ≥18.5 and ≤ 24.9 kg/m2 at screening
* Participant is willing to refrain from consuming alcoholic drinks 24 h prior to test days (V2 - V3)
* Participant is not smoking
* Participant is able and motivated to comply with protocol requirements like for instance take the investigational product the way it is prescribed and to do the tests
* Participant understands the study procedures and signs forms providing informed consent to participate in the study

Exclusion Criteria:

* Participant has abnormal clinical chemistry and haematology laboratory test results of clinical significance that in the judgment of the investigator would interfere with the participant's ability to comply with the study protocol (which might confound the interpretation of the study results), or put the participant at undue risk
* Participants with a history of GI disorders that are likely to interfere with the mode of action of the test product
* Participant has donated more than 300 mL of blood during the three months prior to screening
* Participant has a history, in the judgment of the investigator, of a psychological illness or condition such as to interfere with the participant's ability to understand the requirements of the study
* Use of antibiotics or signs of active systemic infection in the last 6 months
* Participants who are on hypocaloric/hypercaloric diet aiming for weight loss/gain
* Participant has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer
* Participant is pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation
* Regular use of dietary supplements e.g. riboflavin, fish oil, 1 month prior to study inclusion
* Participant has had exposure to any non-registered drug product within 30 days prior to the screening visit
* Recent history of (within 12 months of screening visit) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >60g (men) / 40g (women) pure alcohol per day (1.5 l / 1 l beer resp. 0.75 l / 0.5 l wine)
* Participant has a known allergy or sensitivity to study product or any ingredients of the study product or meals provided
* Use of commercially available probiotic, prebiotic and other supplements that may affect the gut microbiota

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Number of F. prausnitzii per gram faeces | 2 weeks
  To determine the effect of 2 weeks oral riboflavin supplementation (50 and 100 mg/day) on the number of F. prausnitzii per gram faeces in comparison with placebo

SECONDARY OUTCOMES:
Bacterial composition (diversity and quantity of anaerobic microbiota) per gram faeces | 2 weeks
  To determine the effects of 2 weeks oral riboflavin supplementation (50 and 100 mg/day) on bacterial composition (diversity and quantity of anaerobic microbiota) in comparison with placebo
Production of short chain fatty acids (SCFA) in faeces | 2 weeks
  To determine the effects of 2 weeks oral riboflavin supplementation (50 and 100 mg/day) on the production of short chain fatty acids (SCFA) in faeces in comparison with placebo
Gastrointestinal (GI) comfort (bloating, flatulence) | 2 weeks
  To determine the effects of 2 weeks oral riboflavin supplementation (50 and 100 mg/day) on gastrointestinal (GI) comfort (bloating, flatulence) in comparison with placebo using validated visual analogue scale (VAS) questionnaires
Oral Glucose Tolerance Test: blood glucose | 2 weeks
  In a subgroup of participants, to determine the effects of 2 weeks oral riboflavin supplementation (50 and 100 mg/day) on blood glucose, and plasma insulin, GLP-1, GLP-2 and ghrelin as well as appetite feelings during an oral glucose tolerance test (oGTT) in comparison with placebo
Oral Glucose Tolerance Test: plasma insulin | 2 weeks
  In a subgroup of participants, to determine the effects of 2 weeks oral riboflavin supplementation (50 and 100 mg/day) on blood glucose, and plasma insulin, GLP-1, GLP-2 and ghrelin as well as appetite feelings during an oral glucose tolerance test (oGTT) in comparison with placebo
Oral Glucose Tolerance Test: Glucagon-like Peptide 1 (GLP-1) | 2 weeks
  In a subgroup of participants, to determine the effects of 2 weeks oral riboflavin supplementation (50 and 100 mg/day) on blood glucose, and plasma insulin, GLP-1, GLP-2 and ghrelin as well as appetite feelings during an oral glucose tolerance test (oGTT) in comparison with placebo
Oral Glucose Tolerance Test: Glucagon-like Peptide 2 (GLP-2) | 2 weeks
  In a subgroup of participants, to determine the effects of 2 weeks oral riboflavin supplementation (50 and 100 mg/day) on blood glucose, and plasma insulin, GLP-1, GLP-2 and ghrelin as well as appetite feelings during an oral glucose tolerance test (oGTT) in comparison with placebo
Oral Glucose Tolerance Test: ghrelin | 2 weeks
  In a subgroup of participants, to determine the effects of 2 weeks oral riboflavin supplementation (50 and 100 mg/day) on blood glucose, and plasma insulin, GLP-1, GLP-2 and ghrelin as well as appetite feelings during an oral glucose tolerance test (oGTT) in comparison with placebo
Oral Glucose Tolerance Test: Appetite feelings during the test | 2 weeks
  In a subgroup of participants, to determine the effects of 2 weeks oral riboflavin supplementation (50 and 100 mg/day) on blood glucose, and plasma insulin, GLP-1, GLP-2 and ghrelin as well as appetite feelings during an oral glucose tolerance test (oGTT) in comparison with placebo
Changes in stool characteristics: faeces pH | 2 weeks
  To determine the possible changes in stool characteristics such as faeces pH upon riboflavin supplementation
Changes in stool characteristics: dry weight | 2 weeks
  To determine the possible changes in stool characteristics such as dry weight upon riboflavin supplementation
Changes in gut permeability related biomarkers: fatty-acid-binding proteins (I-FABP (plasma)) | 2 weeks
  To determine any possible effect on gut permeability, assessment of permeability related biomarkers: fatty-acid-binding proteins (I-FABP (plasma)) and SM-22 (serum) upon riboflavin supplementation
Changes in gut permeability related biomarkers: SM-22 (serum) | 2 weeks
  To determine any possible effect on gut permeability, assessment of permeability related biomarkers: fatty-acid-binding proteins (I-FABP (plasma)) and SM-22 (serum) upon riboflavin supplementation
Riboflavin concentration in faeces | 2 weeks
  To determine the effects of 2 weeks oral riboflavin supplementation on riboflavin concentration in faeces and plasma
Riboflavin concentration in plasma | 2 weeks
  To determine the effects of 2 weeks oral riboflavin supplementation on riboflavin concentration in faeces and plasma

CONTACTS AND LOCATIONS:
Overall Officials: Hermie J.M. Harmsen, PhD, Principal Investigator — Medical Microbiology UMCG Groningen
Locations (1):
- Medical Microbiology, UMCG Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu L, Sadaghian Sadabad M, Gabarrini G, Lisotto P, von Martels JZH, Wardill HR, Dijkstra G, Steinert RE, Harmsen HJM. Riboflavin Supplementation Promotes Butyrate Production in the Absence of Gross Compositional Changes in the Gut Microbiota. Antioxid Redox Signal. 2023 Feb;38(4-6):282-297. doi: 10.1089/ars.2022.0033. Epub 2022 Oct 10. PMID 35943883